CLINICAL TRIAL: NCT02165046
Title: Randomized, Single-dose, Three-way Crossover Study to Assess the Bioavailability of Using SYN006 HFA MDI (Budesonide/Procaterol 180/10mcg) vs Pulmicort pMDI (Budesonide 200 μg) and Meptin Air (Procaterol 10mcg)" in Healthy Volunteer.
Brief Title: Bioavailability Study of SYN006, Pulmicort pMDI and Meptin Air in Healthy Adult.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intech Biopharm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MCPK09003J1
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Procaterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- SYN006 HFA MDI, 180/10 mcg/dose (Experimental): SYN006 HFA MDI(Budesonide/Procaterol Hydrochloride, 180/10mcg), Single dose, 4 puffs
  Interventions: Drug: Budesonide; Drug: Procaterol
- Pulmicort pMDI (Active Comparator): Budesonide 200mcg, single dose, 4 puffs
  Interventions: Drug: Budesonide
- Meptin Air 10mcg (Active Comparator): Procaterol hydrochloride 10mcg, single dose, 4 puffs
  Interventions: Drug: Procaterol

INTERVENTIONS:
Drug: Budesonide
  Arms: Pulmicort pMDI; SYN006 HFA MDI, 180/10 mcg/dose
Drug: Procaterol
  Arms: Meptin Air 10mcg; SYN006 HFA MDI, 180/10 mcg/dose

SUMMARY:
Budesonide + Procaterol HFA MDI is a novel asthma product containing both budesonide and procaterol in a single inhaler. Budesonide is a corticosteroid that treats underlying airway inflammation in asthma. Procaterol is a direct acting sympathomimetic with predominantly Beta-adrenoceptor stimulant activity selective to Beta-2 receptors (a Beta-2 agonist). It is used as a bronchodilator in the management of reversible airways obstructive pulmonary disease. Budesonide and Procaterol therefore have complementary effects, treating two different components of asthma.

DETAILED DESCRIPTION:
Test drug : SYN006 HFA MDI (Budesonide + Procaterol Hydrochloride) Strength: (Budesonide 180ug and Procaterol Hydrochloride 10ug/puff) Mode of administration: Orally inhaled administration, single dose (4 puffs)

Reference drug 1 : Pulmicort pMDI (Budesonide) Strength: (Budesonide 200ug/puff) Mode of administration: Orally inhaled administration, single dose (4 puffs)

Reference drug 2 : Meptin Air 10ug (Procaterol Hydrochloride) Strength: (Procaterol Hydrochloride 10ug/puff) Mode of administration: Orally inhaled administration, single dose (4 puffs)

One dose for each drug (Test, Reference 1 and Reference 2)with an at least 6-day washout period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision of signed written informed consent before enrollment into the study, ability to communicate with the investigators, and to understand and comply with the requirements of the study.
* 2. Healthy adults, aged between 20 and 40 years old.
* 3. Subjects with Body Mass Index (BMI) of ≧18.5 and ≦25.0 (BMI will be calculated as weight in kilogram [kg]/height in meters2 [m2]).
* 4. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, chest x-ray and electrocardiogram.
* 5. No significant deviation from normal biochemistry examination.
* 6. No significant deviation from normal hematology examination.
* 7. No significant deviation from normal urinalysis examination.

Exclusion Criteria:

* 1. History of drug or alcohol abuse within the past year.
* 2. Medical history of severe drug allergy or sensitivity to analogous drug.
* 3. Evidence of acute or chronic diseases or having undergone surgery from 4 weeks prior to Period I dosing.
* 4. Evidence of any clinical significant renal, cardiovascular, hepatic, hematopoietic, neurological, pulmonary or gastrointestinal pathology.
* 5. Planned vaccination during the time course of the study.
* 6. Taking any clinical investigation drug from 2 months prior to Period I dosing.
* 7. Use of any medication, including herb medicine from 4 weeks before dosing.
* 8. Donation of 500 mL of blood in the past 3 months prior to dosing or donation of 250 mL of blood in the past 2 months prior to dosing.
* 9. A positive Hepatitis B surface antigen or positive Hepatitis C antibody result.
* 10.A positive test for HIV antibody.
* 11.In screening subjects will be given training to ensure that subjects are able to correctly use the investigational products. If the subjects, the use of the investigational products lack of proficiency will not be included in this study.
* 12.Students of National Defense Medical Center.
* 13.For female subjects, if they meet any of the following criteria:

  1. Lactating women
  2. Positive pregnancy test (urine) at screening, or prior to dosing
  3. Do not use adequate contraception during the study
  4. Women taking oral contraceptives

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | predose, 0.083, 0.167, 0.333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 hours post-dose
Maximum plasma concentration (Cmax) | predose, 0.083, 0.167, 0.333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 hours post-dose
Time to reach Maximum plasma concentration (Tmax) | predose, 0.083, 0.167, 0.333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 hours post-dose

SECONDARY OUTCOMES:
Mean residence time (MRT) | predose, 0.083, 0.167, 0.333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 hours post-dose
  To evaluate the safety of the formulations used. The other PK-variables were assessed for description purposes. As safety parameters, adverse events and vital signs (blood pressure, heart rate and body temperature) were recorded.
Plasma elimination rate constant | predose, 0.083, 0.167, 0.333, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14 hours post-dose
  To evaluate the safety of the formulations used. The other PK-variables were assessed for description purposes. As safety parameters, adverse events and vital signs (blood pressure, heart rate and body temperature) were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: C M Perng, M.D, Principal Investigator — Tri-Service General Hospital
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan